CLINICAL TRIAL: NCT04173663
Title: Project ASSIST: Advocating for Supports to Improve Service Transitions
Brief Title: Advocating for Supports to Improve Service Transitions
Acronym: ASSIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: University of Illinois at Urbana-Champaign (Other); University of Wisconsin, Madison (Other)
Responsible Party: Principal Investigator, Julie Taylor, Associate Professor of Pediatrics, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 191187
Record Dates: First submitted 2019-10-09; First posted 2019-11-22 (Actual); Results first posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-12

CONDITIONS: Autism Spectrum Disorder; Autism
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Insemination, Artificial, Heterologous

STUDY DESIGN:
Intervention Model Description: After eligibility is determined and baseline data are collected, parents will be randomized, in two cohorts, to the treatment or materials-only control condition. Given the relatively small sample size in each cohort at each site (n = 30 at each of three sites), simple randomization is not recommended as it might result in unequal group sizes. The investigators will use 1:1 block randomization within each site to give equal number of subjects in each group. To ensure balance of important covariates, the investigators will block on key moderators: whether the youth has an Intellectual Disability (ID) and is in high school. Co-occurring ID and being in vs. out of high school impact service eligibility, and ID impacts the likelihood of post-secondary education (PSE) and community employment. By balancing moderators, the researchers maximize power to detect effect modification of the treatment effect.
Who Masked: Outcomes Assessor
Masking Description: Research personnel collecting follow-up data are masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASSIST intervention group (Experimental): This group will attend the 12 sessions of the ASSIST training program (one 2-hour session per week for 12 weeks).
  Interventions: Behavioral: ASSIST
- Control: Written materials only group (Other): This informational control group will receive the ASSIST binder and all written materials developed for the program on the same schedule as the treatment group but will not attend the group sessions.
  After the treatment group is treated and follow up data is collected for comparison between treatment and control, the control group will have the option to take the ASSIST training program.
  Interventions: Behavioral: ASSIST

INTERVENTIONS:
Behavioral: ASSIST — The ASSIST program is a 12-week advocacy training to educate parents of youth with autism about the adult service system (note that an optional 13th session on secondary transition planning can be offered if ASSIST is being delivered to families of youth who are in high school). It is a group training, comprised of didactic instruction, family-sharing activities, case studies, and group discussions. The ASSIST program for the proposed study will be directed at each site by an experienced Program Facilitator from the community with knowledge about group processes, person-centered planning, and adult service systems, who will be coached by a member of the study team. The ASSIST program will be delivered in full partnership with the local disability community. In most sessions, the Program Facilitator will be aided by community content experts who present the specifics of each topic.

SUMMARY:
This is a randomized intervention study to develop and test the national curriculum of a parent intervention training targeting parent's ability for advocate for services to improve the transition to adulthood for their youth with autism spectrum disorder (ASD).

UPDATE regarding COVID-19: Due to social distancing restrictions, the in-person intervention series that began in Winter 2020 was paused in Spring 2020 for Cohort 1 intervention groups (TN and IL). The series resumed in Summer 2020 via synchronous web-conferencing. In response to continued pandemic regulations, ASSIST was permanently moved to synchronous web-conferencing in Fall 2020, and this method was the mode of delivery for all remaining sessions and series at all sites (TN, IL, WI).

The remaining baseline data was also moved to remote collection through online interview and questionnaires in Spring 2020. The data collection for all follow ups and check ins (6, 12, 18, 24, and 30 month) were completed through web conference and/or phone calls in addition to online surveys. The final data collection for experimental and control groups from all sites will be complete by Summer 2023.

DETAILED DESCRIPTION:
The proposed research plan is designed to develop and test the effectiveness of a national curriculum of the ASSIST (Advocating for SupportS to Improve Service Transition) program, a 12-week parent training program targeting parents' ability to advocate for services to improve the transition to adulthood for youth with autism (note that an optional 13th session on secondary transition planning can be offered if ASSIST is being delivered to families of youth who are in high school).

Preliminary work demonstrated that youth whose parents participated in the "Volunteer Advocacy Program- Transition" or VAP-T (a pilot 12-week intervention program on which ASSIST is based) were more likely to be employed or in postsecondary education (PSE), and received more school-based and adult services, when compared to a wait-list control group.

In the proposed research, the investigators conduct a randomized-controlled trial with 180 families to build on previous findings in four important ways: 1) by making modifications to the program content to make it applicable to service systems across the nation, and rigorously testing whether the ASSIST program is effective when delivered across three states (Tennessee, Illinois, Wisconsin); 2) by incorporating the perspective of offspring with autism into the intervention and data collection; 3) by examining mechanisms by which the ASSIST program influences youth outcomes; and 4) by exploring barriers to participation and factors that moderate treatment response.

The investigators hypothesize that ASSIST participation will improve parents' advocacy ability, leading to higher rates of employment, PSE, social participation, and service access for youth with autism. The investigators will test this hypothesis by randomly assigning parents of transition-aged youth with autism (ages 16-26) to either a treatment or active, materials-only control group, and following families over 3 years. The investigators propose four Specific Aims: (1) To use a multi-site randomized-controlled trial to examine whether ASSIST participation increases parent advocacy ability (i.e. the intervention target); (2) To test whether participating in ASSIST leads to improved youth outcomes (employment, post-secondary education, social participation, service access) during the transition to adulthood; (3) To examine which aspects of parent advocacy ability mediate the relations between ASSIST participation and youth outcomes; and (4) To explore moderators of treatment response and barriers to participation in the intervention.

By rigorously testing a new intervention to improve the transition to adulthood for youth with autism, the proposed research addresses an area of critical need as identified by the 2016-7 Interagency Autism Coordinating Committee Strategic Plan. The project will result in a new intervention to improve outcomes for youth with autism that can be disseminated through state and local agencies across the nation.

ELIGIBILITY:
Inclusion criteria include:

1. parents willing to participate in the ASSIST 12-week intervention, who have an offspring with autism between the ages of 16 and 26 years. This age range was chosen to allow for the testing of whether the ASSIST is more effective if offered prior to versus after high school exit (a key moderator in Aim 4). The investigators set a lower bound of age 16, as that is when transition planning is mandated to have begun in the schools, and an upper bound of age 26 to capture families of youth who are still in the "transition years" as defined by the Institute of Medicine. If both parents in a family want to attend the training, the investigators will allow it but will designate one as the study's primary respondent. There is no minimum or maximum age limit for parent participants.
2. parents are willing to be randomized to the treatment or control condition;
3. parents are able to travel weekly to one of the project sites (Nashville, TN; Chicagoland;IL; Madison/Milwaukee, WI) to participate in the group ASSIST sessions (12 weekly sessions). The responding parent and the offspring with ASD must also be able to travel to a project site for a diagnostic evaluation to confirm the ASD diagnosis (using the gold- standard Autism Diagnostic Observation Schedule-2 or ADOS-2) and to establish IQ and adaptive behavior functioning;
4. the participating parent and youth must live in one of the states where the intervention is being delivered, as the adult service system is different in every state;
5. son/daughter has a previous diagnosis of ASD from an educational or health care provider, and meets lifetime cut-offs for ASD in a telephone screening of the Social Communication Questionnaire. This will decrease the risk that youth fail to meet diagnostic criteria for ASD during the diagnostic evaluation. Note that although the investigators will collect IQ and adaptive behavior information to assess functioning of the offspring with ASD, this information will not be used to determine eligibility; parents of offspring with all levels of functioning can participate in the ASSIST project; and
6. the participating parent is proficient with the English language, as all ASSIST presentations and data collection materials are in English.

Exclusion criteria include:

1. parents unable to participate in the ASSIST 12-week intervention due to scheduling conflicts, or who are unable to travel weekly to one of the sites;
2. parents NOT willing to be randomized to the treatment or control condition;
3. parents and/or youth do NOT live in one of the states where the intervention is being delivered;
4. The youth does not have a previous diagnosis of ASD from an educational or health care provider
5. The youth does not meet lifetime cut-offs for ASD in a telephone screening of the Social Communication Questionnaire, answered by the parent.
6. The participating parent is not proficient with the English language.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2023-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Lounds Taylor, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (3):
- United States (3):
  - University of Illinois at Urbana-Champaign, Chicago, Illinois
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Waisman Center at University of Madison-Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burke,MM, Goldman SE, Hart MS, Hodapp RM. Evaluating the Efficacy of a Special Education Advocacy Training Program: Evaluating the Efficacy of Advocacy Training. Journal of Policy and Practice in Intellectual Disabilities, 13(4), 269-276, 2016.
- [Background] Koren PE, DeChillo N, Friesen, BJ. Measuring empowerment in families whose children have emotional disabilities: A brief questionnaire. Rehabilitation Psychology, 37(4), 305-321, 1992.
- [Background] Sanford C, Newman L, Wagner M, Cameto R, Knokey AM, Shaver D. The Post-High School Outcomes of Young Adults with Disabilities up to 6 Years after High School: Key Findings from the National Longitudinal Transition Study-2 (NLTS2). NCSER 2011-3004. National Center for Special Education Research, 2011.
- [Background] Lounds Taylor J, Adams RE, Bishop SL. Social participation and its relation to internalizing symptoms among youth with autism spectrum disorder as they transition from high school. Autism Res. 2017 Apr;10(4):663-672. doi: 10.1002/aur.1709. Epub 2016 Oct 14. PMID 27739234
- [Background] Taylor JL, Seltzer MM. Developing a vocational index for adults with autism spectrum disorders. J Autism Dev Disord. 2012 Dec;42(12):2669-79. doi: 10.1007/s10803-012-1524-x. PMID 22466690
- [Background] Taylor JL, Hodapp RM, Burke MM, Waitz-Kudla SN, Rabideau C. Training Parents of Youth with Autism Spectrum Disorder to Advocate for Adult Disability Services: Results from a Pilot Randomized Controlled Trial. J Autism Dev Disord. 2017 Mar;47(3):846-857. doi: 10.1007/s10803-016-2994-z. PMID 28070786
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Result] Taylor JL, Pezzimenti F, Burke MM, DaWalt LS, Lee CE, Rabideau C. Development, Feasibility, and Acceptability of a Nationally Relevant Parent Training to Improve Service Access During the Transition to Adulthood for Youth with ASD. J Autism Dev Disord. 2022 Jun;52(6):2388-2399. doi: 10.1007/s10803-021-05128-z. Epub 2021 Jul 7. PMID 34232419
- [Result] Burke MM, Cheung WC, Li C, DaWalt L, Segal J, Taylor JL. Parental Perceptions of Service Access for Transition-Aged Youth With Autism During COVID-19. Intellect Dev Disabil. 2022 Oct 1;60(5):369-381. doi: 10.1352/1934-9556-60.5.369. PMID 36162047
- See also: Transitions Lab Website — https://www.vumc.org/transitionslab

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The data reported only includes parents who were enrolled in the study. Youth did not receive the intervention. For the purposes of primary and secondary outcome measure reporting youth were not considered enrolled and data was not collected
Groups:
- Control: Written Materials Only Group: This informational control group will receive the ASSIST binder and all written materials developed for the program on the same schedule as the treatment group but will not attend the group sessions.
  After the treatment group is treated and follow up data is collected for comparison between treatment and control, the control group will have the option to take the ASSIST training program.
  ASSIST: The ASSIST program is a 12-week advocacy training to educate parents of youth with autism about the adult service system (note that an optional 13th session on secondary transition planning can be offered if ASSIST is being delivered to families of youth who are in high school). It is a group training, comprised of didactic instruction, family-sharing activities, case studies, and group discussions. The ASSIST program for the proposed study will be directed at each site by an experienced Program Facilitator from the community with knowledge about group processes, person-centered planning, and adult service systems, who will be coached by a member of the study team. The ASSIST program will be delivered in full partnership with the local disability community. In most sessions, the Program Facilitator will be aided by community content experts who present the specifics of each topic.
Period: Overall Study
Arm/Group | ASSIST Intervention Group | Control: Written Materials Only Group
Started | 91 | 94
Follow-Up 1 (Intervention-end) | 88 | 88
Follow-Up 2 (6 Month Post-intervention) | 84 | 79
Follow-Up 3 (12 Month Post-intervention) | 81 | 79
Follow-Up 4 (18 Month Post-intervention) | 79 | 75
Follow-Up 5 (24 Month Post-intervention) | 72 | 62
Completed | 73 | 64
Not Completed | 18 | 30
Not completed — Withdrawal by Subject | 1 | 6
Not completed — Lost to Follow-up | 17 | 24

BASELINE CHARACTERISTICS:
Population: The data reported only includes parents who were enrolled in the study. Youth did not receive the intervention. For the purposes of primary and secondary outcome measure reporting youth were not considered enrolled and data was not collected.
Groups:
- Total: Total of all reporting groups
Arm/Group | ASSIST Intervention Group | Control: Written Materials Only Group | Total
Number analyzed (Participants) | 91 | 94 | 185
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 87 | 91 | 178
  >=65 years | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.89 (6.64) | 50.28 (5.91) | 51.07 (6.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 86 | 166
  Male | 11 | 8 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 14
  Not Hispanic or Latino | 84 | 87 | 171
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 7 | 16
  White | 77 | 81 | 158
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 91 | 94 | 185

OUTCOME MEASURES:

1. Primary Outcome: Treatment Target: Change in Parental Empowerment Scale
Description: Examine whether ASSIST participation increases the intervention target of parental empowerment measured using the Family Empowerment Scale (FES). The 34-item questionnaire measures the extent to which parents feel empowered across three dimensions: family, the service system; and the larger community and political environment. Items are rated on a 5-point Likert Scale from 1= not at all true to 5 = very true. The total score can range from 34 to 170, with higher scores indicating greater empowerment.
Time Frame: Baseline to intervention-end, up to month 10
Measure: Mean (Standard Deviation); unit: score on a scale (change score)
Arm/Group | ASSIST Intervention Group | Control: Written Materials Only Group
Number analyzed (Participants) | 88 | 88
score on a scale (change score) | 4.93 (13.72) | 0.61 (14.02)
Statistical Analysis 1: Comparison: ASSIST Intervention Group vs Control: Written Materials Only Group; Test type: Superiority; p = .092, Regression, Linear; Linear regression controlled for study site, cohort, and baseline value of the parental empowerment scale; Slope = -3.27

2. Primary Outcome: Treatment Target: Change in Parental Knowledge About Adult Services Questionnaire
Description: Examine whether ASSIST participation increases the intervention target of parental knowledge about adult service systems. A questionnaire based on a measure developed for the Volunteer Advocacy Program Transition (VAP-T) will be used to evaluate parental knowledge about adult services. The questionnaire consists of 22 multiple-choice questions asking for factual information about adult disability services and the adult disability service system. The total score can range from 0 to 22. Higher scores indicate greater knowledge of the adult disability service system.
Time Frame: Baseline to intervention-end, up to month 10
Population: Of the participants who completed Follow-Up 1, one participant in the intervention group and one person in the control group did not complete this measure, giving us n=87 for the intervention group and n=87 for the control group.
Measure: Mean (Standard Deviation); unit: score on a scale (change score)
Arm/Group | ASSIST Intervention Group | Control: Written Materials Only Group
Number analyzed (Participants) | 87 | 87
score on a scale (change score) | 2.16 (3.00) | 0.20 (2.33)
Statistical Analysis 1: Comparison: ASSIST Intervention Group vs Control: Written Materials Only Group; Test type: Superiority; p = .0000154, Regression, Linear; Linear regression controlled for study site, cohort, and baseline value of the measure; Slope = -1.62

3. Primary Outcome: Treatment Target: Change in Advocacy Skills and Comfort Scale
Description: Examine whether ASSIST participation increases the intervention target of parent advocacy skills measured by the Advocacy Skills and Comfort Scale (ASC). The 10-item measure assesses the degree to which parents feel comfortable and skilled in advocating for their offspring with ASD. Response options range from 1 = not at all to 5 = excellent. The overall score is calculated by averaging all items and can range from 1 to 5, with higher scores indicating more skills/comfort in advocating for their offspring.
Time Frame: Baseline to intervention-end, up to month 10
Measure: Mean (Standard Deviation); unit: score on a scale (change score)
Arm/Group | ASSIST Intervention Group | Control: Written Materials Only Group
Number analyzed (Participants) | 88 | 88
score on a scale (change score) | 0.35 (0.57) | 0.15 (0.55)
Statistical Analysis 1: Comparison: ASSIST Intervention Group vs Control: Written Materials Only Group; Test type: Superiority; p = .014, Regression, Linear; Linear regression controlled for study site, cohort, and baseline value of the measure; Slope = -0.19

4. Primary Outcome: Change in Advocacy Activities Scale
Description: Examine whether ASSIST participation increases the intervention target of parent advocacy activities. The 16-item instrument measures how frequently parents spend time in advocacy activities for the son/daughter with ASD. The response options range from 1 = not at all to 4 = very often. The total score can range from 16 to 64, with higher scores indicating greater parent participation in advocacy activities.
Time Frame: Baseline to 12-month post-intervention, up to month 21
Population: Of the participants who completed Follow-Up 3, eleven participants in the intervention group and three participants in the control group did not complete this measure, giving us n=70 for the intervention group and n=76 for the control group.
Measure: Mean (Standard Deviation); unit: score on a scale (change score)
Arm/Group | ASSIST Intervention Group | Control: Written Materials Only Group
Number analyzed (Participants) | 70 | 76
score on a scale (change score) | -0.84 (6.93) | -1.34 (4.76)
Statistical Analysis 1: Comparison: ASSIST Intervention Group vs Control: Written Materials Only Group; Test type: Superiority; p = 0.883, Regression, Linear; Linear regression controlled for study site, cohort, and baseline value of the measure; Slope = -0.13

5. Primary Outcome: Change in Access to Services Interview: Number of Services the Family Applied for
Description: Test whether parent participation in the ASSIST intervention leads to increase access to services for youth with ASD transitioning from high school to adulthood. Using questions developed for the National Longitudinal Transition Study-2 (NLTS-2), the investigators will collect data (via a semi-structured interview) on the total number of services that the family applied form (e.g., supplemental security income [SSI], vocational rehabilitation services, housing choice voucher). The number of services families can apply for ranges from 0 to 9.
Time Frame: Baseline to 6-month post-intervention, up to month 15; Baseline to 12-month post-intervention, up to month 21
Population: The data analysis only includes parents who were enrolled in the study. Youth did not receive the intervention.
  N reflects the number of participants who completed the measure at each corresponding time point.
Measure: Mean (Standard Deviation); unit: services
Arm/Group | ASSIST Intervention Group | Control: Written Materials Only Group
Number analyzed (Participants) | 83 | 79
services
  Change Score (6 month-Baseline) | 0.07 (0.93) | 0.10 (0.74)
  Change Score (12 month-Baseline): number analyzed (Participants) | 78 | 79
  Change Score (12 month-Baseline) | 0.08 (1.09) | 0.10 (0.76)
Statistical Analysis 1: Comparison: ASSIST Intervention Group vs Control: Written Materials Only Group; Outcome Variable: Number of services family applied for (6 month post intervention); Test type: Superiority; p = .308, Regression, Linear; Linear regression controlled for study site, cohort, and baseline value of the measure; Slope = -0.11
Statistical Analysis 2: Comparison: ASSIST Intervention Group vs Control: Written Materials Only Group; Outcome Variable: Number of services family applied for (12 month post intervention); Test type: Superiority; p = .355, Regression, Linear; Linear regression controlled for study site, cohort, and baseline value of the measure; Slope = -0.11

6. Primary Outcome: Change in Access to Services Interview: Number of Services the Family is Receiving
Description: Test whether parent participation in the ASSIST intervention leads to increase access to services for youth with ASD transitioning from high school to adulthood. Using questions developed for the National Longitudinal Transition Study-2 (NLTS-2) the investigators will collect data (via a semi-structured interview) on total number of services that the family is receiving. For this analysis, services are disaggregated into two types: government (e.g., supplemental security income [SSI], vocational rehabilitation services, housing choice voucher) and direct services (e.g, speech-language pathology, respite care, mental health services). The number of government services the family can receive ranges from 0 to 9. The number of direct services the family can receive ranges from 0 to 21.
Time Frame: Baseline to 6-month post-intervention, up to month 15; Baseline to 12-month post-intervention, up to month 21
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: services
Arm/Group | ASSIST Intervention Group | Control: Written Materials Only Group
Number analyzed (Participants) | 83 | 79
services
  Government Services Change Score (6 month - Baseline) | 0.52 (1.11) | 0.43 (0.90)
  Government Services Change Score (12 month - Baseline): number analyzed (Participants) | 78 | 79
  Government Services Change Score (12 month - Baseline) | 0.50 (1.05) | 0.41 (1.08)
  Direct Services Change Score (6 month - Baseline) | -0.07 (1.87) | -0.33 (2.12)
  Direct Services Change Score (12 month - Baseline): number analyzed (Participants) | 78 | 79
  Direct Services Change Score (12 month - Baseline) | -0.68 (2.05) | -0.37 (2.05)
Statistical Analysis 1: Comparison: ASSIST Intervention Group vs Control: Written Materials Only Group; Outcome Variable: Number of government services family is receiving (6 month post intervention); Test type: Superiority; p = .699, Regression, Linear; Linear regression controlled for study site, cohort, and baseline value of the measure; Slope = -0.06
Statistical Analysis 2: Comparison: ASSIST Intervention Group vs Control: Written Materials Only Group; Outcome Variable: Number of government services the family is receiving (12 month post intervention); Test type: Superiority; p = .573, Regression, Linear; Linear regression controlled for study site, cohort, and baseline value of the measure; Slope = -0.10
Statistical Analysis 3: Comparison: ASSIST Intervention Group vs Control: Written Materials Only Group; Outcome Variable: Number of direct services the family is receiving (6 month post intervention); Test type: Superiority; p = .430, Regression, Linear; Linear regression controlled for study site, cohort, and baseline value of the measure; Slope = -0.23
Statistical Analysis 4: Comparison: ASSIST Intervention Group vs Control: Written Materials Only Group; Outcome Variable: Number of direct services the family is receiving (12 month post intervention); Test type: Superiority; p = .391, Regression, Linear; Linear regression controlled for study site, cohort, and baseline value of the measure; Slope = 0.27

7. Primary Outcome: Post-Secondary Youth Outcomes
Description: Test whether parent participation in the ASSIST intervention leads to increase in post-secondary vocational and educational participation for youth with ASD. The Vocational Index will be used to gather information on employment and post-secondary educational programs that youth with ASD are attending / attended 6 months after the intervention. The Vocational Index will be administered via structured interview. This measure is only applicable to youth who have exited high school.
Time Frame: Baseline to 6-month post-intervention, up to month 15; Baseline to 12-month post-intervention, up to month 21
Population: The number analyzed reflects the number of participants who completed the measure at each corresponding time point.
Measure: Count of Participants; unit: Participants
Arm/Group | ASSIST Intervention Group | Control: Written Materials Only Group
Number analyzed (Participants) | 31 | 30
Participants
  Number of participants who had no activities at baseline but activities at 6 month post intervention | 7 | 4
  Number of participants who had no activities at baseline but activities at 12month post intervention: number analyzed (Participants) | 29 | 29
  Number of participants who had no activities at baseline but activities at 12month post intervention | 2 | 5
Statistical Analysis 1: Comparison: ASSIST Intervention Group vs Control: Written Materials Only Group; Outcome Variable: Whether participants were engaged or not engaged in vocational/educational activities (6 month post intervention); Test type: Superiority; p = .510, Regression, Logistic; Logistic regression controlled for study site, cohort, and baseline value of the measure; Slope = -0.44
Statistical Analysis 2: Comparison: ASSIST Intervention Group vs Control: Written Materials Only Group; Outcome Variable: Whether participants were engaged or not engaged in vocational/educational activities (12 month post intervention); Test type: Superiority; p = .296, Regression, Logistic; Logistic regression controlled for study site, cohort, and baseline value of the measure; Slope = 0.64

8. Secondary Outcome: Social Participation Youth Outcomes
Description: Test whether parent participation in the ASSIST intervention leads to increase in social participation for youth with ASD. Questions developed to measure social participation will be used to measure the social participation achievements of the youth participants before and after ASSIST per parent-report. This measure consists of 10 items with a 5-point Likert scale ranging from 0 = Less than yearly or never to 4 = Several times a week. The total score can range from 0 to 40, with higher scores indicating greater social participation for the youth with ASD.
Time Frame: Baseline to 12-month post-intervention, up to month 21
Population: Of the participants who completed Follow-Up 3, twelve participants in the intervention group and eight participants in the control group did not complete this measure, giving us n=69 for the intervention group and n=71 for the control group.
Measure: Mean (Standard Deviation); unit: score on a scale (change score)
Arm/Group | ASSIST Intervention Group | Control: Written Materials Only Group
Number analyzed (Participants) | 69 | 71
score on a scale (change score) | 0.13 (4.38) | -0.72 (4.78)
Statistical Analysis 1: Comparison: ASSIST Intervention Group vs Control: Written Materials Only Group; Test type: Superiority; p = .361, Regression, Linear; Linear regression controlled for study site, cohort, and baseline value of the measure; Slope = -0.66

9. Secondary Outcome: Change in Access to Services Interview: Unmet Service Needs
Description: Test whether parent participation in the ASSIST intervention leads to decrease in unmet service needs for youth with ASD transitioning from high school to adulthood. Using questions developed for the National Longitudinal Transition Study-2 (NLTS-2), the investigators will collect data (via a semi-structured interview) on total number of unmet service needs that the family is experiencing / experienced.
Time Frame: Baseline to 6-month post-intervention, up to month 15; Baseline to 12-month post-intervention, up to month 21
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: unmet needs
Arm/Group | ASSIST Intervention Group | Control: Written Materials Only Group
Number analyzed (Participants) | 83 | 79
unmet needs
  Change Score (6 month - Baseline) | -0.28 (2.54) | -0.43 (2.37)
  Change Score (12 month - Baseline): number analyzed (Participants) | 78 | 79
  Change Score (12 month - Baseline) | -0.35 (2.59) | -0.70 (2.38)
Statistical Analysis 1: Comparison: ASSIST Intervention Group vs Control: Written Materials Only Group; Outcome Variable: Number of unmet service needs (6 month post intervention); Test type: Superiority; p = .810, Regression, Linear; Linear regression controlled for study site, cohort, and baseline value of the measure; Slope = -0.08
Statistical Analysis 2: Comparison: ASSIST Intervention Group vs Control: Written Materials Only Group; Outcome Variable: Number of unmet service needs (12 month post intervention); Test type: Superiority; p = .678, Regression, Linear; Linear regression controlled for study site, cohort, and baseline value of the measure; Slope = -0.13

10. Secondary Outcome: Access to Services Interview: Barriers to Service Receipt
Description: Test whether parent participation in the ASSIST intervention is associated with fewer barriers to services for youth with ASD transitioning from high school to adulthood. Using questions developed for the National Longitudinal Transition Study-2 (NLTS-2), the investigators will collect data (via a semi-structured interview) on the number of barriers to services experienced.
Time Frame: Baseline to 12-month post-intervention, up to month 21
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: barriers
Arm/Group | ASSIST Intervention Group | Control: Written Materials Only Group
Number analyzed (Participants) | 70 | 76
barriers | 2.66 (2.03) | 2.71 (1.91)
Statistical Analysis 1: Comparison: ASSIST Intervention Group vs Control: Written Materials Only Group; Test type: Superiority; p = .924, Regression, Linear; Linear regression controlled for study site and cohort,; Slope = 0.03

ADVERSE EVENTS:
Time Frame: 36 months
Arm/Group | ASSIST Intervention Group | Control: Written Materials Only Group
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/94
Serious Adverse Events (participants affected / at risk) | 0/91 | 0/94
Other Adverse Events (participants affected / at risk) | 17/91 | 17/94
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASSIST Intervention Group (N=91) | Control: Written Materials Only Group (N=94)
Unanticipated Problem (Social circumstances) | 17 (17) | 17 (17) — Breech in confidentiality that may involve risk. Study team member emailed 34 participants utilizing cc rather than bcc which allowed email addressed to be shared. This was not related to intervention. This was related to data collection.

LIMITATIONS AND CAVEATS:
We could not analyze whether treatment targets mediate the relationship between ASSIST participation and youth outcomes of employment/PSE, social participation, and service access (specific aim 3), as we did not detect a treatment effect.

The results of the trial were likely impacted by the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-08-10): https://cdn.clinicaltrials.gov/large-docs/63/NCT04173663/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT04173663/SAP_001.pdf
  • Informed Consent Form (2019-10-04): https://cdn.clinicaltrials.gov/large-docs/63/NCT04173663/ICF_002.pdf